CLINICAL TRIAL: NCT00436592
Title: Safety and Efficacy of NeuroFlo in 8-24 Hour Stroke Patients
Acronym: Flo 24
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CoAxia (Industry)
Responsible Party: Flo 24 Steering Committee, CoAxia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0240
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Cerebrovascular Accident
Keywords: acute; ischemic; stroke; device; treatment
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: NeuroFlo™ Catheter

INTERVENTIONS:
Device: NeuroFlo™ Catheter — 45 minute Treatment

SUMMARY:
The purpose of this study is to assess the safety and feasibility of the NeuroFlo™ catheter in treating patients with ischemic stroke whose last time symptom-free was between 8-24 hours prior to treatment. The NeuroFlo device is intended to increase blood flow to the brain and potentially reduce the damage caused by stroke.

DETAILED DESCRIPTION:
The study is a prospective, single arm treatment feasibility trial to determine the baseline safety and feasibility of the NeuroFlo device in acute ischemic stroke patients whose last known time symptom-free is between 8-24 hours.

A maximum of 25 patients at 5 US sites and 25 patients at 10 Canadian & European sites may be enrolled in this initial study phase. An independent data safety and monitoring board will assess the safety of the treatment on a routine basis.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* NIHSS between 4-20
* Time from symptom onset between 8 and 24 hours

Exclusion Criteria:

* Hemorrhagic stroke
* Certain types of heart disease
* Kidney disease
* Other conditions the doctor will assess

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Assessment of all adverse events from baseline to 30 days post-treatment. | 30 Days

SECONDARY OUTCOMES:
Potential benefit will be assessed through collection of neurological indices at baseline, post-procedure, 24 hours, day 4 (or discharge), 30 and 90 days. | 90 Days
Cerebral perfusion changes associated with device therapy will be assessed using MRI perfusion studies acquired at baseline and ≤ 4 hours post-procedure. | ≤ 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Flo 24 Steering Committee, Study Chair — Multiple Organizations
Locations (10):
- United States (5):
  - UCLA, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
- Germany (2):
  - University of Erlangen, Erlangen
  - University of Essen, Essen
- CHUV Lausanne, Lausanne, Switzerland

REFERENCES:
- [Derived] Hammer MD, Schwamm L, Starkman S, Schellinger PD, Jovin T, Nogueira R, Burgin WS, Sen S, Diener HC, Watson T, Michel P, Shuaib A, Dillon W, Liebeskind DS. Safety and feasibility of NeuroFlo use in eight- to 24-hour ischemic stroke patients. Int J Stroke. 2012 Dec;7(8):655-61. doi: 10.1111/j.1747-4949.2011.00719.x. Epub 2012 Jan 20. PMID 22264202
- See also: Related Info — http://www.coaxia.com